CLINICAL TRIAL: NCT00155090
Title: Proton Magnetic Resonance Spectroscopy of Normal Breast Tissues in Women Volunteers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700788
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-01

CONDITIONS: Breast Neoplasms
Keywords: Magnetic resonance imaging,; breast disease
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Magnetic resonance spectroscopy (MRS) is a diagnostic technique in MRI that distinguishes various metabolites on the basis of their slightly different chemical shifts or resonance frequencies. The Proton is the most abundant nucleus in the body. We will try to establish the typical proton MRS pattern of normal women breasts to be a guideline for future further investigations.

DETAILED DESCRIPTION:
There are few reports regarding proton MRS in normal female breasts. The fibroglandular tissues and fat are the two major gross components in the breast. The water content in the fibroglandular tissues is much higher than that in the fat. There is still no documented report discussing proton MRS in normal female breasts of premenopausal and postmenopausal women. Our study is to evaluate the proton MRS findings among normal premenopausal and postmenopausal women breasts, to find out if there are statistical differences on the main proton MRS patterns, water and lipid peak intensities and ratios between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* women age ranged 30 years of age or older, with normal mammograms or ultrasound in recent 3 months

Exclusion Criteria:

* any women not fulfilling the inclusion criteria

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Jane Wang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Kvistad KA, Bakken IJ, Gribbestad IS, Ehrnholm B, Lundgren S, Fjosne HE, Haraldseth O. Characterization of neoplastic and normal human breast tissues with in vivo (1)H MR spectroscopy. J Magn Reson Imaging. 1999 Aug;10(2):159-64. doi: 10.1002/(sici)1522-2586(199908)10:23.0.co;2-0. PMID 10441019